CLINICAL TRIAL: NCT00003803
Title: A Randomized Phase III Study Comparing Induction Chemotherapy to Daily Low Dose Cisplatin Both Combined With High Dose Radiotherapy Using Concomitant Boost Technique in Patients With Inoperable Non-Small Cell Lung Cancer Stage I, II, and Low Volume Stage III
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Stage I, Stage II, or Stage III Non-small Cell Lung Cancer That Cannot Be Surgically Removed
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-08972-22973; EORTC-08972
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage III non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy used high-energy x-rays to damage tumor cells. It is not yet know whether chemotherapy followed by radiation therapy is more effective than chemotherapy given with radiation therapy for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of chemotherapy and radiation therapy in treating patients who have unresectable stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare survival, disease-free survival, local control, and pattern of recurrence in patients with unresectable stage I, II, or low-volume stage III non-small lung cancer treated with high-dose radiotherapy either preceded by induction chemotherapy with gemcitabine and cisplatin or combined with daily cisplatin.
* Compare the acute and late toxic effects of these regimens in these patients.
* Determine the quality of life of these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to performance status (0 vs 1), TNM stage, and participating center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and cisplatin IV over 3-6 hours on day 2. Treatment is repeated once 21 days later. Patients undergo high-dose accelerated conformal radiotherapy beginning on week 9 (day 57), 5 days a week, for 24 fractions, using a concurrent boost technique up to 66 Gy.
* Arm II: Patients receive low-dose cisplatin IV followed 1-2 hours later by high-dose accelerated conformal radiotherapy. Treatment continues daily, 5 days a week, for 24 fractions, using a concurrent boost technique up to 66 Gy.

Quality of life is assessed before treatment and at weeks 9-11, 19, 27, and 35.

Patients are followed at 3 weeks, 6-7 weeks, and then every 8 weeks thereafter.

PROJECTED ACCRUAL: A total of 418 patients (209 per arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage I, II, III (T1-4, N0-3, M0)

    * No metastases to supraclavicular, contralateral hilar, or contralateral scalene lymph nodes
  * Medically inoperable or unresectable
* No pleural or pericardial effusion (except with repeated negative cytology)

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 6.8 g/dL
* No hemoptysis causing a decrease of hemoglobin of 1 g/dL or more within 24 hours

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.25 times normal OR
* Creatinine clearance greater than 70 mL/min

Cardiovascular:

* No evidence of heart failure
* No myocardial infarction within the past 6 months
* No superior vena cava syndrome

Pulmonary:

* FEV1 at least 1 L
* No pre-existing fibrotic lung disease
* No postobstructive pneumonia preventing exact delineation of tumor volume
* Diffusion capacity at least 60%

Other:

* No weight loss of more than 10% in the past 3 months
* No uncontrolled infection
* No serious medical risk factors involving any of the major organ systems that would preclude adherence to the study treatment schedule

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the chest
* Maximum length of the esophagus receiving 40 Gy no greater than 18 cm
* Maximum length of the esophagus receiving 66 Gy no greater than 12 cm
* Must limit the spinal cord dose to a maximum of 50 Gy
* Must be able to exclude 25% of the heart from the boost volume

Surgery:

* Not specified

Other:

* No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 1999-02; Primary Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Belderbos, MD, Study Chair — The Netherlands Cancer Institute
Locations (17):
- Belgium (2):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Hopital de Jolimont, Haine-Saint-Paul
- CHR de Grenoble - La Tronche, Grenoble, France
- Mutterhaus der Borromaerinnen, Trier, Germany
- Netherlands (12):
  - Medisch Centrum Haaglanden, 's-Gravenhage (Den Haag, the Hague)
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen - Lokatie Lukas, Apeldoorn
  - Amphia Ziekenhuis, Breda
  - Amphia Ziekenhuis - locatie Molengracht, Breda
  - Reinier de Graaf Group, Delft
  - Radiotherapeutisch Instituut-(Riso), Deventer
  - Catharina Ziekenhuis, Eindhoven
  - Twee Steden Ziekenhuis Vestiging Tilburg, Tilburg
  - Dr. Bernard Verbeeten Instituut, Tilburg
  - Sophia Ziekehuis, Zwolle
- Western General Hospital, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Result] Belderbos J, Uitterhoeve L, van Zandwijk N, Belderbos H, Rodrigus P, van de Vaart P, Price A, van Walree N, Legrand C, Dussenne S, Bartelink H, Giaccone G, Koning C; EORTC LCG and RT Group. Randomised trial of sequential versus concurrent chemo-radiotherapy in patients with inoperable non-small cell lung cancer (EORTC 08972-22973). Eur J Cancer. 2007 Jan;43(1):114-21. doi: 10.1016/j.ejca.2006.09.005. Epub 2006 Nov 3. PMID 17084621